CLINICAL TRIAL: NCT05902182
Title: A Prospective, Multi Centre, Interventional, Non-comparator, Open Label Post Market Clinical Follow up Study to Demonstrate the Efficacy and Safety of Convatec ConvaFoam™ Silicone, ConvaFoam™ Border and ConvaFoam™ Non-adhesive Dressings to Protect Against Skin Breakdown
Brief Title: Study to Demonstrate the Efficacy and Safety of Convatec ConvaFoam™ Silicone, ConvaFoam™ Border and ConvaFoam™ Non-adhesive Dressings to Protect Against Skin Breakdown
Acronym: DONNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WC-22-426
Record Dates: First submitted 2023-04-28; First posted 2023-06-13 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2023-08

CONDITIONS: Skin Breakdown

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ConvaFoam Dressings (Experimental): All participants skin areas will be assessed and allocated a dressing based upon the investigator's clinical judgement. They will receive either ConvaFoam Border, Silicone or Non-Adhesive for up to 2 weeks as an addition to their standard pressure injury prevention protocol.
  Interventions: Device: ConvaFoam

INTERVENTIONS:
Device: ConvaFoam — ConvaFoam™ Silicone, ConvaFoam™ Border and ConvaFoam™ non-adhesive dressings are designed to provide a moist wound healing environment and removing dead-space between the wound and dressing interface. These dressings are designed to manage excess exudate levels which may further damage the wound bed and surrounding skin. In addition, the dressings are designed to protect fragile skin from moisture, shear, and friction damage. These will be used in line with the patients pressure injury mitigation protocol for a 2 week period, with daily inspections of the skin area.

SUMMARY:
A prospective, multi centre, interventional, non-comparator, open label study to demonstrate the efficacy, safety, and performance of ConvaFoam™ Silicone, ConvaFoam™ Border and ConvaFoam™ Non-adhesive to protect against skin breakdown

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over
* Patients able and willing to provide informed consent/Personal Consultee/Nominated consultee/ Their nominated consultee
* Intact healthy skin
* Stage I pressure ulcer/injury
* Patients who are at risk of developing skin breakdown (injury), in any clinical setting, with at least one clinically vulnerable area (including but not limited to sacrum, heel, elbows, hips, ischial tuberosity and spine)
* Braden score of 12 or less

Exclusion Criteria:

* Patients with known allergies to any of the materials used in the dressing
* Subjects requiring any oxidising agents such as hydrogen peroxide or hypochlorite solutions
* Patients who are at high risk of unavoidable skin breakdown for example caused by a medical device (for example, under ventilation or faecal management systems)
* Patients with a wound of any aetiology on the area under investigation Patients who, in the opinion of the investigator, are considered unsuitable for any other reason
* Patients with a history of previous healed pressure ulcer/ injury in the area under investigation
* Patients who demonstrate a deterioration of skin from baseline skin assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To measure the efficacy of ConvaFoam™ Silicone, ConvaFoam™ Border and ConvaFoam™ non-adhesive dressings when used to protect of skin against breakdown. | 2 weeks
  This will be measured by:
  • The incidence of skin breakdown

SECONDARY OUTCOMES:
To assess the safety of ConvaFoam™ Silicone, ConvaFoam™ Border and ConvaFoam™ non-adhesive dressings when used to protect skin against breakdown. | 2 weeks
  This will be measured via reporting all device related adverse events and device malfunctions, such as allergic reactions, bleeding, pain/discomfort in area of dressing, skin irritation, and reported as per protocol
To assess the performance of ConvaFoam™ Silicone, ConvaFoam™ Border and ConvaFoam™ non-adhesive dressings when used to protect skin against breakdown. | 2 weeks
  This will be measured by reporting:
  The number of times the dressing has been lifted and reapplied before needing to be replaced compared to the instructions for use. The ability of the dressing to be reapplied to the skin following skin assessments as per the patients standard of care.

IPD SHARING:
Plan to Share IPD: No